CLINICAL TRIAL: NCT00781703
Title: DIAMOND Study: Evaluation of a Natural Experiment to Improve Statewide Depression Care in MN
Brief Title: Evaluation of a Natural Experiment to Improve Statewide Depression Care in Minnesota (MN)
Acronym: DIAMOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: PAR-06-039; R01MH080692 (NIH)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- DIAMOND Care Model (Other): Patients in activated clinic sites will receive the DIAMOND depression care model, including a care manager, frequent use of the Patient Health Questionnaire-9 (PHQ9), treatment adjustment as indicated, psychiatric consultation, relapse prevention.
  Interventions: Other: DIAMOND depression care model

INTERVENTIONS:
Other: DIAMOND depression care model — Patients in activated clinic sites will receive the DIAMOND depression care model, including a care manager, frequent use of the PHQ9, treatment adjustment as indicated, psychiatric consultation, relapse prevention.

SUMMARY:
The study will evaluate a unique natural experiment that aims to transform the primary care of patients with depression. The experiment's aim is to cause statewide implementation of an evidence-based care model for depression by changing the reimbursement system and by using an established regional collaborative (the Institute for Clinical Systems Improvement) to both facilitate the model's widespread use and certify that medical groups have implemented it. Study hypotheses include the following:

1. Newly treated depressed patients in medical groups that have implemented the new reimbursement and facilitation will report receiving higher rates of best care processes than such patients in these medical groups before implementation.
2. Rates of best care practices reported to be received by newly treated depressed patients two years after each medical group implements changes will be maintained at least at the rate reported by patients one year post implementation.
3. Newly treated depressed patients in medical groups that have participated in the new reimbursement and facilitation will have greater improvement in depression symptoms and work productivity and lower healthcare costs than such patients in groups before participation.
4. Medical group measures of priority for improving depression care, capability to manage change, and practice systems will be predictive of more patient-reported best care processes, both at one point in time and in change over time.

DETAILED DESCRIPTION:
The study will use a multiple baseline across settings with staggered implementation to test the effects of changed reimbursement and facilitated organizational change on the use and sustainability of evidenced-based care processes for patients with depression. The study will also test the effect of the care process changes on changes in depression symptoms, healthcare costs, and work productivity.

ELIGIBILITY:
Inclusion Criteria:

* major depression
* Patient Health Questionaire (PHQ-9) > 9
* primary care management of depression

Exclusion Criteria:

* comorbid psychiatric conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2631 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Rates of best care processes | baseline, 6 months

SECONDARY OUTCOMES:
Improvement in depression symptoms, work productivity and total healthcare costs | baseline, 3 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Leif I Solberg, MD, Principal Investigator — HealthPartners Institute